CLINICAL TRIAL: NCT06843447
Title: A Phase 1b/2 Open-label, Multicenter Study to Evaluate the Safety and Efficacy of Raludotatug Deruxtecan With or Without Other Anticancer Investigational Agents in Participants With High-grade Serous Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer Who Have Relapsed After Prior Platinum-based Chemotherapy
Brief Title: A Clinical Study of Raludotatug Deruxtecan in People With Ovarian Cancer (MK-5909-003)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5909-003; MK-5909-003 (Other: MSD); 2024-514674-47-00 (Registry Identifier: EU CT); U1111-1308-2821 (Registry Identifier: UTN); REJOICE-Ovarian02 (Other: MSD)
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer Recurrent
MeSH Terms: interventions — Carboplatin; Paclitaxel; Bevacizumab; pembrolizumab

STUDY DESIGN:
Masking Description: This is an open-label study; therefore, the Sponsor, investigator, and participant will know the intervention administered.
  Imaging data will be centrally reviewed by independent radiologist(s) without knowledge of participant dose assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort A-1 Arm 1 (R-DXd + Carboplatin Dose 1) (Experimental): Participants receive escalating doses of intravenous (IV) raludotatug deruxtecan in combination with carboplatin at Dose 1. Participants can receive up to a maximum of six 3-week cycles of carboplatin (approximately 4 months) and will receive raludotatug deruxtecan until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Drug: Carboplatin; Drug: Rescue Medication
- Cohort A-1 Arm 2 (R-DXd + Paclitaxel) (Experimental): Participants receive escalating doses of IV raludotatug deruxtecan in combination with paclitaxel. Participants can receive up to a maximum of six 3-week cycles of paclitaxel (approximately 4 months) and will receive raludotatug deruxtecan until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Drug: Paclitaxel; Drug: Rescue Medication
- Cohort A-1 Arm 3 (R-DXd + Carboplatin Dose 2) (Experimental): Participants receive escalating doses of intravenous (IV) raludotatug deruxtecan in combination with carboplatin at Dose 2. Participants can receive up to a maximum of six 3-week cycles of carboplatin (approximately 4 months) and will receive raludotatug deruxtecan until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Drug: Carboplatin; Drug: Rescue Medication
- Cohort B-1 (R-DXd + Bevacizumab) (Experimental): Participants receive escalating doses of IV raludotatug deruxtecan in combination with bevacizumab until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Biological: Bevacizumab; Drug: Rescue Medication
- Cohort B-2 (R-DXd Phase 2 + Bevacizumab) (Experimental): Participants with platinum-resistant recurrent ovarian cancer (PRROC) receive recommended Phase 2 dose (RP2D) of IV raludotatug deruxtecan in combination with bevacizumab until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Biological: Bevacizumab; Drug: Rescue Medication
- Cohort C-1 (R-DXd + Pembrolizumab) (Experimental): Participants receive escalating doses of IV raludotatug deruxtecan in combination with pembrolizumab. Participants can receive up to a maximum of thirty-five 3-week cycles of pembrolizumab (approximately 2 years) and will receive raludotatug deruxtecan until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Drug: Rescue Medication; Biological: Pembrolizumab
- Cohort D (R-DXd Phase 2 +/- Bevacizumab) (Experimental): Participants with platinum-sensitive recurrent ovarian cancer (PSROC) receive RP2D of IV raludotatug deruxtecan in combination with or without bevacizumab until disease progression or discontinuation.
  Interventions: Biological: Raludotatug Deruxtecan; Biological: Bevacizumab; Drug: Rescue Medication

INTERVENTIONS:
Biological: Raludotatug Deruxtecan — IV infusion on Day 1 of every 3-week cycle.
  Other Names: MK-5909, R-DXd
Drug: Carboplatin — IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles.
  Arms: Cohort A-1 Arm 1 (R-DXd + Carboplatin Dose 1); Cohort A-1 Arm 3 (R-DXd + Carboplatin Dose 2)
Drug: Paclitaxel — IV infusion on Day 1 of every 3-week cycle for a maximum of 6 cycles.
  Arms: Cohort A-1 Arm 2 (R-DXd + Paclitaxel)
Biological: Bevacizumab — IV infusion on Day 1 of every 3-week cycle.
  Other Names: Includes, based on sourcing:; - Avastin®; - Alymsys®; - MVASI®; - Oyavas®; - Zirabev®; - Vegzelma®; - Aybintio®; - Breztri®
  Arms: Cohort B-1 (R-DXd + Bevacizumab); Cohort B-2 (R-DXd Phase 2 + Bevacizumab); Cohort D (R-DXd Phase 2 +/- Bevacizumab)
Drug: Rescue Medication — Includes 5-HT3 Serotonin Receptor Antagonist, NK-1 receptor antagonist, and corticosteroid, administered per protocol.
Biological: Pembrolizumab — IV infusion on Day 1 of every 3-week cycle for a maximum of 35 cycles.
  Arms: Cohort C-1 (R-DXd + Pembrolizumab)

SUMMARY:
Researchers are looking for other ways to treat relapsed high-grade serous ovarian cancer. Relapsed means the cancer came back after treatment. High-grade means the cancer cells grow and spread quickly. Serous means the cancer started in the cells that cover the ovaries, the lining of the belly, or in the fallopian tubes.

Standard treatment (usual treatment) for people with relapsed high-grade serous ovarian cancer may include:

* Chemotherapy, which is a treatment that uses medicine to destroy cancer cells or stop them from growing
* Targeted therapy, which is a treatment that works to control how specific types of cancer cells grow and spread

Raludotatug deruxtecan (R-DXd) is a study treatment that is an antibody drug conjugate (ADC). An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells. Researchers want to know if R-DXd is safe to take with other treatments and if people tolerate them together. They also want to learn how many people have the cancer respond (gets smaller or goes away) to the treatments.

DETAILED DESCRIPTION:
This study has 2 parts: Part 1 is a dose escalation phase of R-DXd. Part 2 is the efficacy expansion phase and will use the Recommended Phase 2 Dose (RP2D) of R-DXd determined in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Has pathologically documented diagnosis of high-grade serous epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* Has measurable disease per Response Evaluation Criteria In Solid Tumors 1.1
* Participants in Cohort A-1 Arm 2 and Arm 3: Has relapsed disease after 1 to 3 prior lines of therapy and radiographic evidence of disease progression ≥6 months (≥180 days) after the last dose of platinum-based therapy (ie, platinum-sensitive disease).
* Participants in Cohort B-1 and Cohort B-2: Has relapsed disease after 1 to 3 prior lines of therapy and radiographic evidence of disease progression <6 months (<180 days) after the last dose of platinum-based therapy (ie, platinum-resistant disease).
* Participants in Cohort B-1 and Cohort B-2: Is a candidate for bevacizumab treatment
* Has provided tumor tissue from a core or excisional biopsy of a tumor lesion not previously irradiated
* Has an Eastern Cooperative Oncology Group performance status of 0 to 1 assessed within 7 days before allocation
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy
* Participants who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load prior to allocation
* Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Participants in Cohort C-1 and Cohort D: Has relapsed disease after 1 prior line of therapy, radiographic evidence of disease progression ≥6 months (≥180 days) after the last dose of platinum-based therapy (ie, platinum-sensitive disease) and progressed during prior treatment with PARPi in the first-line setting

Exclusion Criteria:

* Has any of the following within 6 months before allocation: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event
* Has uncontrolled or significant cardiovascular disease
* Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, and any autoimmune, connective tissue, or inflammatory disorders with potential pulmonary involvement, or prior pneumonectomy
* Has ≥Grade 2 peripheral neuropathy
* Has received prior treatment with cadherin-6-targeted agents
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks or 5 half-lives (whichever is shorter) before allocation
* Has received prior radiotherapy within 2 weeks of the start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Receives chronic steroid treatment
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active CNS metastases and/or carcinomatous meningitis
* Has history of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD
* Has active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-03-27 (Estimated); Study Completion 2029-03-27 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experience a Dose-limiting Toxicity (DLT) Per Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE v5.0) | Up to 21 days
  DLTs are defined as toxicities during the DLT evaluation period that are assessed by the investigator to be possibly, probably, or definitely related to study treatment and include: Grade 4 thrombocytopenia of any duration or Grade 3 thrombocytopenia lasting ≥7 days; Grade 3 or higher thrombocytopenia associated with clinically significant bleeding; Grade 4 lymphocytopenia lasting ≥14 days; Grade 4 anemia of any duration; any other Grade 4 hematologic toxicity lasting ≥7 days; febrile neutropenia Grade 3 or Grade 4 meeting pre-specifications; pre-specified hepatic organ toxicities; all Grade 3 or higher other nonhematologic toxicities except those pre-specified; other pre-specified nonhematologic toxicities; any delay in treatment with the planned dose of ≥21 days or discontinuation of treatment due to a toxicity during the DLT evaluation period, or Grade 5 toxicity. The number of participants with DLTs will be reported.
Part 1: Number of Participants with One or More Adverse Events (AEs) | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants with one or more AEs will be reported.
Part 1: Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.
Part 2: Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Part 1: Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants who have a confirmed Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumours version 1.1 (RECIST 1.1). ORR will be assessed by blinded independent central review (BICR).
Part 2: Duration of Response (DOR) | Up to approximately 3 years
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by Blinded Independent Central Review (BICR) will be presented.
Part 2: Progression-free Survival (PFS) | Up to approximately 3 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Part 2: Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from the first dose of study treatment to death due to any cause.
Part 2: Number of Participants with One or More AEs | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.
Part 2: Number of Participants who Discontinue Study Intervention Due to an AE | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (16):
- United States (5):
  - The University of Louisville, James Graham Brown Cancer Center ( Site 0009), Louisville, Kentucky
  - Memorial Sloan Kettering Cancer Center ( Site 0003), New York, New York
  - Houston Methodist Hospital ( Site 0010), Houston, Texas
  - START Mountain Region ( Site 0008), West Valley City, Utah
  - University of Virginia Health System ( Site 0011), Charlottesville, Virginia
- Israel (3):
  - Rambam Health Care Campus ( Site 0202), Haifa
  - Shaare Zedek Medical Center ( Site 0201), Jerusalem
  - Sheba Medical Center ( Site 0200), Ramat Gan
- Spain (5):
  - Institut Català d'Oncologia - L'Hospitalet ( Site 0302), L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra ( Site 0301), Madrid, Madrid, Comunidad de
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0300), Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-START Madrid-FJD ( Site 0303), Madrid
  - Hospital Universitario 12 de Octubre ( Site 0304), Madrid
- United Kingdom (3):
  - Royal Marsden Hospital ( Site 0402), Fulham, England
  - The Royal Marsden NHS Foundation Trust. ( Site 0403), Sutton, England
  - Barts Health NHS Trust ( Site 0401), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com